CLINICAL TRIAL: NCT03006497
Title: The Efficacy of Exercise Program Based on Motor Learning Principles in Correction of Forward Head Posture
Brief Title: Exercise Program Based on Motor Learning and Forward Head Posture Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eleni Kapreli (Other)
Responsible Party: Sponsor-Investigator, Eleni Kapreli, Associate Professor, Physiotherapy Department, Technological Education Institute of Sterea Ellada
Organization: Technological Education Institute of Sterea Ellada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHYSMSC1
Record Dates: First submitted 2016-12-03; First posted 2016-12-30 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Musculoskeletal Abnormalities; Deformity
Keywords: neck; motor control; motor learning
MeSH Terms: conditions — Musculoskeletal Abnormalities; Congenital Abnormalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will not participate in any exercise program. However, at the end, home based exercises and special advice will be given to the participants.
- Intervention (Experimental): The intervention group will participate in an exercise program based on motor learning principles for 4 weeks/3 sessions per week, for a total of 12 sessions of 30-45 minutes each.
  Interventions: Other: Exercise program based on motor learning principles

INTERVENTIONS:
Other: Exercise program based on motor learning principles — The exercise program will include simple activities exposing volunteers in various environmental conditions with a view to adjust their head posture in such conditions. The progressiveness of exercises will be based on the two-dimensional classification system of Gentile (1987). Furthermore, external attentional focus will be used.
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate the efficiency of an exercise program based on principles of motor learning in correction of Forward Head Position (FHP) in asymptomatic patients.

DETAILED DESCRIPTION:
Epidemiological studies have shown that bad posture and poor body control occurs at puberty, with forward head posture (FHP) and rounded shoulders being the most common biomechanical deviations in sagittal plane. The FHP is defined as an anterior displacement of the head with hyperextension of the cervical spine and this is associated with a reduction in the length of the upper portion of the trapezius, posterior portion of the cervical extensor muscles, the sternocleidomastoid and the levator scapulae. FHP can be evaluated by measuring craniovertebral angle (CVA) which is defined as the angle between a horizontal line passing through C7 and a line extending from the tragus of the ear to C7.

CVA, smaller than 50 degrees, constitute a criterion of abnormal posture of cervical spine, suggesting FHP. People with FHP present incomplete balance control, thereby affecting the position of the center of gravity and motor control of the body. The establishment of altered motor control strategies could lead to balance disorders, neck muscle imbalances, chronic neck pain and even respiratory dysfunction.

Despite the efforts of researchers to create effective treatment programs based on strength training and stretching exercises, positive long-term results have been a problem in FHP correction. For this reason, re-education of posture and body alignment, through exercise programs based on motor learning, with cognitive elements (attention, motivation, feedback, reasoning), could be proved a more effective therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Students at Technological Educational Institute of Sterea Ellada,
* Aged 18-26 years old
* Males and females
* Craniocervical angle < 50 degrees (statical Forward Head Posture in standing position)

Exclusion Criteria:

* Injury or surgery in cervical spine
* Accompanying neurologic, musculoskeletal or mental problems
* Any medical administration
* Intense continuous or intermittent neck pain
* BMI >25
* Participation in any rehabilitation or physiotherapy sessions considering neck dysfunction the last 6 months
* Change in physical activities during the research period of 6 weeks

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01; Primary Completion 2017-05 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Static Forward Head Posture (sFHP) | Change from Baseline sFHP at 4 weeks and Change from Baseline sFHP at 6 weeks
  The sFHP will be assessed by calculating the craniovertebral angle through lateral photographs in standing. The craniovertebral angle is the angle between the line extending from the tragus of the ear to the 7th cervical vertebra (C7) spinous process and the horizontal line through C7. The calculation of the angle on the photographs will be carried out using AutoCAD software. A performance curve will be developed using the measurements during the 4 weeks practice and 2 weeks after the end of protocol (retension test).
Change of Dynamic Forward Head Posture (dFHP) | Change from Baseline dFHP t at 4 weeks and Change from Baseline dFHP at 6 weeks
  The dFHP will be assessed by calculating the craniovertebral angle through video motion during walking. The craniovertebral angle is the angle between the line extending from the tragus of the ear to the 7th cervical vertebra (C7) spinous process and the horizontal line through C7. The calculation of the angle The calculation of the angle will be carried out using Kinovea and AutoCAD softwares. dFHP will be regarded as a transfer test. Transfer tests are tests involving some novel situation, so that people must adapt the skill they have been practicing to the characteristics of this new situation.

SECONDARY OUTCOMES:
Overall self-esteem | Baseline; week 4; week 6
  Sorensen self-esteem test will be used which has been translated into Greek and has been tested for its reliability and validity.
Mood | Baseline; week 4; week 6
  A ten point Visual Analogue Scale (VAS) will be used
Overall physical fatigue | Baseline; week 4; week 6
  A ten point VAS scale will be used
Overall mental fatigue | Baseline; week 4; week 6
  A ten point VAS scale will be used
Attention-concentration | Baseline; week 4; week 6
  Attention- concentration questionnaire will be used. It has been developed in Greek language and has been tested for its reliability and validity.
Verbal Comprehension index | Baseline
  The Wechsler Adult Intelligence Scale (WAIS-IV) (similarities) will be used. Participants will be given a number of pairs of words or concepts and have to describe how they are similar.
Perceptual Organization Index | Baseline
  The WAIS-IV (Matrix Reasoning) will be used. Participants will be given pictures of sets of drawings and have to choose the correct drawing that is missing from each set.
Change in Deep neck flexors endurance | Change from Baseline Deep neck flexors endurance at 4 weeks and Change from Baseline Deep neck flexors endurance at 6 weeks
  The first stage of the test allows for the quantification of the performance of craniocervical flexion action, while the second stage examines the isometric endurance of deep neck flexors, during which the participant adopts the crook lying position. The air chamber of a pressure biofeedback device is positioned under the cervical area and the participant is asked to perform a head nod action at five different pressure levels (22, 24, 26, 28 and 30 mmHg). The test is initially performed at a pressure level of 22 mmHg and proceeds to the next pressure level if the participant is able to maintain in the position for 10 seconds on three separate occasions. The Chattanooga stabilizer pressure biofeedback will be used.
Change in Discomfort | Change from Baseline discomfort at 4 weeks and Change from Baseline discomfort at 6 weeks
  The Discomfort will be assessed using a ten point grade VAS scale, where 0 is no pain and 10 worst pain.
Change in Area of Discomfort | Change from Baseline discomfort at 4 weeks and Change from Baseline discomfort at 6 weeks
  The Discomfort (Head, Neck, Shoulders and upper arms, Middle back, Lower back, Forearms and Wrists/hands areas) will be assessed using a body chart
Weight | Baseline
  Measurement of weight with scale (kilograms)
Height | Baseline
  Measurement of height (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Eleni V Kapreli, MSc, PhD, Study Chair — Technological Educational Institute of Sterea Ellada; Stefani Argyrou, BSc, Principal Investigator — Technological Educational Institute of Sterea Ellada

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) are to be shared with other researchers, when it will be available

REFERENCES:
- [Background] Christakou A, Zervas Y, Psychountaki M, Stavrou NA. Development and validation of the attention questionnaire of rehabilitated athletes returning to competition. Psychol Health Med. 2012;17(4):499-510. doi: 10.1080/13548506.2011.630402. Epub 2011 Nov 25. PMID 22114988
- [Background] Dimitriadis Z, Kapreli E, Strimpakos N, Oldham J. Respiratory weakness in patients with chronic neck pain. Man Ther. 2013 Jun;18(3):248-53. doi: 10.1016/j.math.2012.10.014. Epub 2012 Nov 28. PMID 23199797
- [Background] Dimitriadis Z, Kapreli E, Strimpakos N, Oldham J. Reliability of the chin tuck neck flexion test for assessing endurance of short neck flexors in healthy individuals. Physiother Theory Pract. 2015 May;31(4):299-302. doi: 10.3109/09593985.2014.1002874. Epub 2015 Jan 14. PMID 25585517
- [Background] Han J, Park S, Kim Y, Choi Y, Lyu H. Effects of forward head posture on forced vital capacity and respiratory muscles activity. J Phys Ther Sci. 2016 Jan;28(1):128-31. doi: 10.1589/jpts.28.128. Epub 2016 Jan 30. PMID 26957743
- [Background] Kang JH, Park RY, Lee SJ, Kim JY, Yoon SR, Jung KI. The effect of the forward head posture on postural balance in long time computer based worker. Ann Rehabil Med. 2012 Feb;36(1):98-104. doi: 10.5535/arm.2012.36.1.98. Epub 2012 Feb 29. PMID 22506241
- [Background] Kapreli E, Vourazanis E, Strimpakos N. Neck pain causes respiratory dysfunction. Med Hypotheses. 2008;70(5):1009-13. doi: 10.1016/j.mehy.2007.07.050. Epub 2007 Oct 23. PMID 17959320
- [Background] Rosario JL, Diogenes MS, Mattei R, Leite JR. Can sadness alter posture? J Bodyw Mov Ther. 2013 Jul;17(3):328-31. doi: 10.1016/j.jbmt.2012.12.001. Epub 2012 Dec 23. PMID 23768277
- [Background] Ruivo RM, Carita AI, Pezarat-Correia P. The effects of training and detraining after an 8 month resistance and stretching training program on forward head and protracted shoulder postures in adolescents: Randomised controlled study. Man Ther. 2016 Feb;21:76-82. doi: 10.1016/j.math.2015.05.001. Epub 2015 May 13. PMID 26028408
- [Background] Silva AG, Johnson MI. Does forward head posture affect postural control in human healthy volunteers? Gait Posture. 2013 Jun;38(2):352-3. doi: 10.1016/j.gaitpost.2012.11.014. Epub 2012 Dec 7. PMID 23219786
- [Background] Wulf G, Mercer J, McNevin N, Guadagnoli MA. Reciprocal influences of attentional focus on postural and suprapostural task performance. J Mot Behav. 2004 Jun;36(2):189-99. doi: 10.3200/JMBR.36.2.189-199. PMID 15130869